CLINICAL TRIAL: NCT05431582
Title: Phase I Study of ZN-c3 and Bevacizumab ± Pembrolizumab in Metastatic CCNE1 Amplified and TP53 Mutant Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Zentalis Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0175; NCI-2022-05251 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-02

CONDITIONS: Tumors; Ovarian Cancer; Breast Cancer; Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms | interventions — Bevacizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (Experimental): ZN-c3 in combination with bevacizumab
  Interventions: Drug: ZN-c3; Drug: Bevacizumab
- Regimen B (Experimental): ZN-c3 in combination with bevacizumab and pembrolizumab
  Interventions: Drug: ZN-c3; Drug: Bevacizumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ZN-c3 — Given by PO 1 time a day with a glass (about 8 ounces) of water
Drug: Bevacizumab — Given by vein over about 30-60 minutes on Day 1 of each cycle
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Pembrolizumab — Given by vein over 30-60 minutes on Day 1 of each cycle.
  Other Names: KEYTRUDA®
  Arms: Regimen B

SUMMARY:
Primary Objectives are to determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of ZN-c3 and ZN-c3 and bevacizumab or ZN-c3 and bevacizumab plus pembrolizumab in metastatic CCNE1 amplified and TP53 mutant solid tumors as well to evaluate antitumor activity of ZN-c3 and bevacizumab or ZN-c3 and bevacizumab plus pembrolizumab in metastatic CCNE1 amplified and TP53 mutant solid tumors.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of ZN-c3 and ZN-c3 and bevacizumab or ZN-c3 and bevacizumab plus pembrolizumab in metastatic CCNE1 amplified and TP53 mutant solid tumors.
* To evaluate antitumor activity of ZN-c3 and bevacizumab or ZN-c3 and bevacizumab plus pembrolizumab in metastatic CCNE1 amplified and TP53 mutant solid tumors.

Secondary Objectives:

* To assess progression-free survival (PFS), overall survival (OS), and duration of response (DOR)
* To explore potential biomarkers.
* To explore patient reported outcomes (PRO).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed metastatic solid tumors harboring CCNE1 amplification and TP53 mutation pre-identified in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory, either refractory to standard therapy or for which no effective standard therapy that increases survival for at least 3 months is available, or they declined standard of care therapy.
2. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
3. Male or female aged ≥18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

   Adequate organ functions as defined below:

   Absolute neutrophil count (ANC) ≥ 1,500 /μL. Hemoglobin (Hb) ≥ 8 g/dL. Platelets ≥ 100,000 /μL. Total bilirubin ≤ 1.5 x upper limit of normal (ULN); or total bilirubin < 3.0 x ULN with direct bilirubin ≤ ULN in patients with well documented Gilbert's Syndrome.

   ALT ≤ 3 ULN or ≤ 5 ULN if liver metastases persist. Serum albumin ≥ 3 g/dL. Urinalysis ≤ 1 proteinuria, or urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g.

   PT/INR or partial thromboplastin time (PTT) test < 1.3 the laboratory ULN if not on therapeutic anticoagulation.

   Calculated creatinine clearance (CrCl) ≥ 60 mL/min by the Cockcroft-Gault method* or 24-hour urine collection.

   * CrCl = (140-age) x (weight/kg) x Fa / (72 x serum creatinine mg/dL). a where F= 0.85 for females and F=1 for male
5. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to initiation of therapy (C1D1), and must agree to use effective birth control during the study prior to the first dose and for at least 6 months after the last dose (or longer based on local requirements). Female patients are not considered to be of child-bearing potential if they are post-menopausal (no menses for 12 months without an alternative medical cause) or permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy). Male patients must agree to abstain or use barrier contraception (i.e. condoms), and avoid sperm donation for the duration of the study and for 6 months after treatment stops.
6. Ability to read and fully understand the requirements of the trial, willingness to comply with all trial visits and assessments, and willingness and ability to sign an institutional review board (IRB)-approved written informed consent document (ICD). Patients with Impaired Decision Making Capacity (IDMC) must have a close caregiver or Legally Authorized Representative (LAR).
7. Any prior palliative radiation must have been completed at least 14 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment (Radiotherapy for extended field within 4 weeks or limited field radiotherapy within 2 weeks).
8. Fridericia's corrected QT interval (QTcF =QT/∛(60/HR) ) ≤ 460 milliseconds (ms) for males and ≤ 480 ms for females on ECG conducted at rest during Screening.

   Note: Patients with an atrioventricular pacemaker or other condition (for example, right bundle branch block) that renders the QT measurement invalid are an exception and this criterion does not apply.
9. Ability to take oral medications without medical history of malabsorption or other chronic gastrointestinal disease, or other conditions that may hamper compliance and/or absorption of the study agents. Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN).
10. Provision of an archival tissue block, or 10 formalin-fixed paraffin-embedded (FFPE) slides, or fresh tumor biopsy.
11. Prior treatment with VEGF inhibition or immunotherapy is allowed. But prior treatment with Wee1 kinase inhibition is not allowed.

Exclusion Criteria:

1. Any treatment specifically for systemic tumor control given within 3 weeks before the initiation of therapy; within 2 weeks if cytotoxic agents were given weekly, within 6 weeks for nitrosoureas or mitomycin C; within 5 half-lives for targeted agents with half-lives and pharmacodynamic effects lasting < 5 days; or failure to recover from toxic effects of any previous therapy. A drug that has not received regulatory approval for any indication within 14 or 21 days of treatment for a non-myelosuppressive or myelosuppressive agent, respectively: patients must recover for previous cancer therapy, and are ready to proceed with further cancer therapy.
2. Uncontrolled intercurrent illness including but not limited to:

   * ongoing or active infection requiring intravenous antibiotics
   * symptomatic congestive heart failure (New York Heart Association Class III or IV)
   * history of myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months before study enrollment
   * lesions invading or encasing any major blood vessels and cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
   * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment
   * history or current evidence of uncontrolled ventricular arrhythmia
   * congenital long QT syndrome, or any known history of torsade de pointes, or family history of unexplained sudden death
   * clinically significant bleeding or active gastric or duodenal ulcer
   * chronic diarrhea diseases considered to be clinically significant
   * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment, or any gastrointestinal disorders associated with a high risk of perforation or fistula formation.
   * other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.

   Note: Subjects with a diagnosis of incidental, subsegmental pulmonary embolism or deep vein thrombosis are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment.
3. Unresolved clinically significant Grade 1 or higher toxicity from prior therapy.
4. History of allergic reactions to the study drugs, or any component of the products.
5. Presence of other active invasive cancers that do not harbor CCNE1 amplification and TP53 mutation and requires active treatment other than hormonal therapy.
6. Having not recovered from a major surgical procedure or significant traumatic injury (i.e., still needing additional surgical or medical care for these issues): major surgical procedures ≤ 28 days of treatment entry, or minor surgical procedures ≤ 7 days. No waiting period required following port-a-cath or other central venous access placement. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
7. Currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study. If a patient is currently enrolled in a clinical trial involving non-approved use of a therapeutic device for cancer control, then agreement with the investigator and the sponsor is required to establish eligibility.
8. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: Bacille Calmette-Guérin vaccine, measles, mumps, rabies, rubella, typhoid vaccine, varicella/zoster, and yellow fever. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed.
9. Received strong inhibitors and inducers and sensitive substrates of CYP3A4, as well as strong and moderate p-glycoprotein (P-gp) inhibitors (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers), which cannot be discontinued within 2 weeks of the initiation of study therapy, withheld during the study until 2 weeks after the last dose of study drug.
10. Symptomatic primary tumors or metastasis in the brain and/or central nervous system that are uncontrolled with antiepileptics and/or require steroids at a dose of prednisone > 10 mg/day or equivalent.
11. Evidence of leptomeningeal or lymphangitic carcinomatosis.
12. A history of another primary malignancy that is currently clinically significant, requiring active intervention except for hormone therapy.
13. Lactation or pregnancy.
14. Human immunodeficiency virus requiring HAART treatment due to unknown drug-drug interactions or has known history of active hepatitis B or C. However, patients with history of active hepatitis B or C are eligible if their hepatitis is well controlled. Screening tests for HIV, HBV and HCB are not mandatory.

    Individuals must not meet these additional criteria if they participate in the study to receive the pembrolizumab-based combination regimen:
15. Concurrent immunosuppressive therapy or steroid (> 10 mg/day prednisone or equivalent).
16. History of autoimmune disease including but not limited to inflammatory bowel disease, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, which requires systemic therapy in the past 2 years.

    Note: Patients with vitiligo, resolved childhood asthma/atopy, hypothyroidism on stable hormone replacement, controlled asthma, Type I diabetes, Graves' disease, or Hashimoto's disease, are not excluded.
17. History of grade ≥ 3 immune-related adverse events with previous immunotherapy. Note: Patients with adequately treated skin rash other than Steven-Johnson, toxic epidermal necrolysis of other severe forms of dermatitis; or replacement therapy for endocrinopathies, are not excluded.
18. History of interstitial lung disease or (non-infectious) pneumonitis that required steroids or current pneumonitis.
19. History of grade ≥ 3 allergic reaction to treatment with a monoclonal antibody.
20. Anti-PD-(L)1 naïve patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of ZN-c3 . | through study completion, an average of 1 year
To establish the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) ZN-c3 and bevacizumab. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org